CLINICAL TRIAL: NCT06603857
Title: A Prospective, Placebo-controlled, Double-blinded, Randomized Clinical Trial Evaluating the Efficacy and Tolerability of Pre and Post Care Skincare Regimen Paired With 1927nm Diode Fractional Laser for Photodamage on the Face
Brief Title: Skin Care Regimen for Improving Photoaging Signs on the Face
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: L'Oreal (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Skinceuticals CE Ferulic 2024
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Improve Photoaging Signs
Keywords: wrinkles; aging; photodamage

STUDY DESIGN:
Intervention Model Description: Prospective, placebo-controlled, double-blinded, randomized study
Who Masked: Outcomes Assessor
Masking Description: The blinded investigator will perform assessments at all study visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): Subjects who will receive two treatments with 1927nm (Clear and Brilliant Perméa®) non-ablative fractional diode laser for rejuvenation of photodamaged skin of the face in pairing with Skinceuticals CE Ferulic
  Interventions: Drug: CE Ferulic; Device: 1927nm (Clear and Brilliant Perméa®)
- Group B (Sham Comparator): Subjects who will receive two treatments with 1927nm (Clear and Brilliant Perméa®) non-ablative fractional diode laser for rejuvenation of photodamaged skin of the face in pairing with vehicle serum
  Interventions: Drug: Sham Comparator; Device: 1927nm (Clear and Brilliant Perméa®)

INTERVENTIONS:
Drug: CE Ferulic — CE Ferulic serum regimen combined with laser treatment
  Arms: Group A
Drug: Sham Comparator — Vehicle serum regimen combined with laser treatment
  Arms: Group B
Device: 1927nm (Clear and Brilliant Perméa®) — non-ablative fractional diode laser

SUMMARY:
Compare the effectiveness of laser treatment using CE Ferulic versus vehicle pre/post laser.

DETAILED DESCRIPTION:
Evaluate the efficacy and tolerability of a Skinceuticals CE Ferulic® when used once daily over the course of 14 weeks with 2-week pre-treatment period and 12-week treatment period in pairing with two pre-elected laser treatments with 1927nm non-ablative fractional diode laser treatment for improving skin photoaging signs on the face.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 30-70 years (Fitzpatrick I-IV 30-65 years, Fitzpatrick V-VI 30-70 years)
* Fitzpatrick skin types I-VI
* Subjects in good general health based on investigator's judgment and medical history
* Must be willing to give and sign an informed consent form and photographic release form
* Must be willing to have examinations of face and digital photographs performed of the face
* Physician evaluator classifying the subject as mild to moderate (Score 3-6) on the modified Griffiths 10-Point Scale for the face.
* The subject must be planning to undergo fractional non-ablative laser resurfacing to the face and bilateral postauricular area and be willing to comply with study protocol and complete the entire course of the study.
* Subjects using any treatment skincare products (per investigator discretion) must discontinue use of these products four weeks before the start of participating in this clinical study and for the duration of the study.
* Male subjects with facial hair must be willing to shave prior to every visit.
* Must be willing to maintain usual sun exposure
* Subject agrees to avoid tanning or use of sunless tanner during the entire course of the study
* Negative urine pregnancy test result at the time of study entry (if applicable)
* For female subjects of childbearing potential, must be willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment.
* A female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation.
* Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants, Implanon®, Depo-Provera®, double-barrier methods (e.g., condoms and spermicide), abstinence, and/or vasectomy of partner with a documented second acceptable method of birth control, should the subject become sexually active.
* Must be willing to comply with study treatments and complete the entire course of the study

Exclusion Criteria:

* Energy-based device (i.e., radiofrequency device treatments, microfocused ultrasound device or other ultrasound-based device treatments, laser and light-based device treatments, microneedling) treatment in the treatment area in the last 6 months
* Chemical peel or microdermabrasion of the face within 60 days prior to enrollment in the study
* Dermal fillers, biostimulators, or neurotoxins treatments of the face during the 6-month period before the study period or planning to undergo during the study period
* Surgery (i.e., face lift, eyebrow lift, neck lift or lower rhytidectomy, liposuction to the neck and/or submentum, etc.) during the 12-month period before study treatment
* Any investigational treatment for improvement of skin quality and/or photodamage of facial skin during the 6-month period before the study treatment
* Use of topical steroids, tretinoin, adapalene, tazarotene, hydroquinone, imiquimod, 5-fluorouracil, ingenol mebutate, concentrated hydrogen peroxide, diclofenac, or photodynamic therapy (PDT) to the face within the previous 4 weeks
* Subjects must not currently be taking isotretinoin (Accutane).
* Creams/cosmeceuticals and/or home therapies to prevent or treat photodamage, uneven skin pigmentation, excessive erythema (redness), fine lines/wrinkles, skin laxity and/or pore size during the 4-week period before study treatment
* Subjects with scarring in the treatment areas
* Subjects with tattoos in the treatment areas
* Subjects with a significant history or current evidence of a medical, psychological, or other disorder that, in the investigator's opinion, would preclude enrollment into the study
* Subjects with a history of or presence of any skin condition/disease (including but not limited to any visible rash, atopic dermatitis, psoriasis, actinic keratoses, keratinocyte carcinoma, melanoma, etc.) in the treatment area that might interfere with the diagnosis or evaluation of study parameters
* Skin with open wounds, excessively sensitive skin, neurotic excoriations, dermatitis or inflammatory rosacea in the treatment area
* History of keloid or hypertrophic scarring
* Subjects with an active bacterial, viral, or fungal infection of the treatment areas or systemic infection
* Subjects who spray tanned or used sunless tanners in the treatment areas four (4) weeks prior to study treatment
* History of lidocaine and/or tetracaine sensitivity deemed by the investigator to preclude the subject from enrolling into the study
* Individuals with known allergies or sensitivities to any of the ingredients of any topical or injectable products being used in this study
* Subjects must not have a compromised ability for wound healing, such as:

malnutrition, steroid use, history of collagen vascular disease (e.g., lupus, scleroderma), atopic dermatitis, or immunologic abnormalities such as vitiligo.

* Subjects planning any cosmetic procedure to the treatment areas during the study period, other than the treatment that will be performed by the investigator
* Presence of incompletely healed wound(s) in the treatment area
* Subjects who are on an immunosuppressant or have an autoimmune condition
* Female subjects who are pregnant, planning a pregnancy, or breast feeding during the study
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-27 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Global Fine Lines | Screening, Baseline, Day 28, Day 56, Day 84
  Score 0 thru 9
  Score 0= No fine lines present; skin looks completely smooth Score 9= Numerous, many fine lines densely packed together in the treatment area
Overall Hyperpigmentation/ Discoloration | Screening, Baseline, Day 28, Day 56, Day 84
  Score 0 thru 9
  Score 0= No hyperpigmentation Score 9= Significant hyperpigmentation, numerous spots, uneven skin tone
Skin Tone Evenness | Screening, Baseline, Day 28, Day 56, Day 84
  Score 0 thru 9
  Score 0= Very even tone Score 9= Uneven, discolored appearance (brown and/or red colors)
Skin Elasticity | Screening, Baseline, Day 28, Day 56, Day 84
  Score 0 thru 9
  Score 0= Skin feels toned, dense Score 9= Skin feels pliable, thin and non-resilient
Skin Firmness | Screening, Baseline, Day 28, Day 56, Day 84
  Score 0 thru 9
  Score 0= Firm, tight feeling skin Score 9= Loose, lax feeling skin
Skin Radiance/ Brightness | Screening, Baseline, Day 28, Day 56, Day 84
  Score 0 thru 9
  Score 0= Very radiant, luminous or glowing appearance Score 9= Very dull/ matte and/or sallow skin appearance
Skin Texture Smoothness | Screening, Baseline, Day 28, Day 56, Day 84
  Score 0 thru 9
  Score 0= Very smooth, even-looking skin texture, no roughness Score 9= Very rough, pronounced, extensive visible skin roughness
Global Wrinkles | Screening, Baseline, Day 28, Day 56, Day 84
  Score 0 thru 9
  Score 0= No wrinkles present, no visible deep, wide and long wrinkles, skin looks smooth Score 9= Numerous wrinkles, deep, wide and long, densely packed together in the treatment area

SECONDARY OUTCOMES:
Tolerability Assessment | Baseline, Day 28
  Stinging/Burning:
  None No stinging/burning of the treatment area Mild Slight, but definite burning of the treatment area Moderate Definite stinging/burning of the treatment area Severe Marked stinging/burning of the treatment area
  Itching:
  None No itching of the treatment area Mild Slight, but definite itching of the treatment area Moderate Definite itching of the treatment area Severe Marked itching of the treatment area
  Rash:
  None No new rash over the treatment area Mild New rash covering some of the treatment area Moderate New rash covering much of the treatment area Severe New rash covering the entirety of the treatment area
  Tightness:
  None No tightness of the treatment area Mild Slight, but definite tightness of the treatment area Moderate Definite tightness of the treatment area Severe Marked tightness of the treatment area
Dermatology Quality of Life Index (Page 1) | Screening, Baseline, Day 28, Day 56, Day 84
  1. Over the last week, how itchy, sore, painful or stinging has your skin been:
     Very Much A lot A little Not at all
  2. Over the last week, how embarrassed or self-conscious have you been because of your skin:
     Very Much A lot A little Not at all
  3. Over the last week, how much has your skin interfered with you going shopping or looking after your home or garden:
     Very Much A lot A little Not at all
  4. Over the last week, how much has your skin influenced the clothes you wear:
     Very Much A lot A little Not at all
  5. Over the last week, how itchy, sore, painful or stinging has your skin been:
     Very Much A lot A little Not at all
  6. Over the last week, how much has your skin made it difficult for you to do any sport:
  Very Much A lot A little Not at all
Dermatology Quality of Life Index (Page 2) | Screening, Baseline, Day 28, Day 56, Day 84
  7.Over the last week, has your skin prevented you from working or studying: Yes or No 7a. If "no", over the last week how much has your skin been a problem at work or studying: Very Much A lot A little Not at all
  8.Over the last week, how much has your skin created problems with your partner or any of your close friends or relatives: Very Much A lot A little Not at all
  9.Over the last week, how much has your skin caused any sexual difficulties: Very Much A lot A little Not at all
  10.Over the last week, how much of a problem has the treatment for your skin been, for example by making your home messy, or by taking up time: Very Much A lot A little Not at all
Subject Self-Assessment Questionnaire (Page 1) | Screening, Baseline, Day 28, Day 56, Day 84
  1. Skin feels more comfortable:
     Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  2. Skin appears younger looking:
     Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  3. Skin appears healthier:
     Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  4. Skin looks renewed/ revitalized:
     Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  5. Skin looks firmer:
     Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  6. Skin feels elastic:
     Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  7. Redness looks reduced:
  Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
Subject Self-Assessment Questionnaire (Page 2) | Screening, Baseline, Day 28, Day 56, Day 84
  8. With the product I'm more satisfied with the procedure results: Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  9. The product reduced the downtime of the procedure or makes the downtime more acceptable: Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  10. The product improves the outcome of the procedure: Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  11. With this product, I would feel more confident to do another procedure: Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  12. I would recommend this product post-procedure: Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
Subject Self-Assessment Questionnaire (Page 3) | Screening, Baseline, Day 28, Day 56, Day 84
  13. It's the best post-procedure care I've ever used (if relevant) : Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  14. It is something I would use after future laser treatments: Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  15. The product has a pleasant texture: Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  16. The product absorbs quickly in to the skin: Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  17. It is a product I would recommend to others: Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly

CONTACTS AND LOCATIONS:
Locations (1):
- West Dermatology Research Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No